CLINICAL TRIAL: NCT05744349
Title: Percutaneous Intramedullary K-wires Fixation of Pediatric Shaft Both Bone Forearm Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Hamdy Abdelmajeed, Resident at the department of Orthopedic surgery and Traumatology Sohag University Hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-02-01
Record Dates: First submitted 2023-02-15; First posted 2023-02-27 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Fracture Fixation, Intramedullary; Fracture Forearm

STUDY DESIGN:
Intervention Model Description: After administration of anesthesia, surgery will be performed with the patient supine on the operating table and fracture will be analyzed with an image intensifier. In radius, the wire will be inserted by surgical drilling through Lister's tubercle or the radial styloid while in ulna, the wire will be inserted through the tip of the olecranon.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients who are younger than the age of 10 years old from both genders and suffering from displaced fractures of shaft both bone of the forearm
  Interventions: Procedure: K-wires Fixation of Pediatric Shaft Both Bone Forearm Fractures

INTERVENTIONS:
Procedure: K-wires Fixation of Pediatric Shaft Both Bone Forearm Fractures — After administration of anesthesia, surgery will be performed with the patient supine on the operating table and fracture will be analyzed with an image intensifier. In radius, the wire will be inserted by surgical drilling through Lister's tubercle or the radial styloid while in ulna, the wire will be inserted through the tip of the olecranon.

SUMMARY:
This study is to improving outcome of pediatric both bone forearm fractures using minimally invasive procedure by intramedullary K-wires.

DETAILED DESCRIPTION:
Most shaft injuries present no unusual challenges and require nothing more than skillful closed reduction and cast immobilization due to the unique property of the growth potential of the immature skeleton. There is a relatively high incidence of re-displacement, malunion and consequent limitation of movement. Perfect anatomical reduction is not always necessary since remodeling of malunion may correct any residual deformity. Angulation has been shown to affect the range of pronation and supination of the forearm.

The most common indications for surgery are failure of closed reduction, open fractures, and fracture instability. When operative intervention is indicated different techniques can be employed such as intramedullary nailing, osteosynthesis with plate and screws fixation and external fixators. Intramedullary nailing has been shown to produce excellent clinical results and in contrast to plate fixation is considered as a minimal invasive procedure.

Surgical technique of K-wires :

After administration of anesthesia, surgery will be performed with the patient supine on the operating table and fracture will be analyzed with an image intensifier. In radius, the wire will be inserted by surgical drilling through Lister's tubercle or the radial styloid while in ulna, the wire will be inserted through the tip of the olecranon.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are younger than the age of 10 years old from both genders and suffering from displaced fractures of shaft both bone of the forearm;
2. Standard preoperative anteroposterior (AP) and lateral forearm radiographs;
3. Complete clinical and radiographic data.

Exclusion Criteria:

1. Poly-traumatized patients with other associated fractures;
2. Undisplaced fractures;
3. Open fractures;
4. Pathological fractures;
5. Malignancy;
6. Malnutrition;
7. Chronic diseases as renal, hepatic, cardiac patients;
8. Incomplete radiographic data.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Union of fractures | 1 month
Degree of flexion and extension at wrist joint | 3 months
Degree of supination and pronation | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yong B, Yuan Z, Li J, Li Y, Southern EP, Canavese F, Xu H. Single Bone Fixation versus Both Bone Fixation for Pediatric Unstable Forearm Fractures: A Systematic Review and Metaanalysis. Indian J Orthop. 2018 Sep-Oct;52(5):529-535. doi: 10.4103/ortho.IJOrtho_125_17. PMID 30237611
- [Background] Cruz AI Jr, DeFroda SF, Gil JA, Hansen H, Bolous A, Procaccini M, Zonfrillo MR. Patient and Parent Satisfaction With Sling Use After Pediatric Upper Extremity Fractures: A Randomized Controlled Trial of a Customized Cast-Sling Versus Standard Cast and Sling. J Pediatr Orthop. 2019 Feb;39(2):e120-e124. doi: 10.1097/BPO.0000000000001091. PMID 29049268
- [Background] Pesenti S, Litzelmann E, Kahil M, Mallet C, Jehanno P, Mercier JC, Ilharreborde B, Mazda K. Feasibility of a reduction protocol in the emergency department for diaphyseal forearm fractures in children. Orthop Traumatol Surg Res. 2015 Sep;101(5):597-600. doi: 10.1016/j.otsr.2015.06.003. Epub 2015 Jul 18. PMID 26198018
- [Background] Sinikumpu JJ, Lautamo A, Pokka T, Serlo W. The increasing incidence of paediatric diaphyseal both-bone forearm fractures and their internal fixation during the last decade. Injury. 2012 Mar;43(3):362-6. doi: 10.1016/j.injury.2011.11.006. Epub 2011 Dec 6. PMID 22154046